CLINICAL TRIAL: NCT05704972
Title: Investigation of Risk Factors Encountered by Operating Room Nurses
Acronym: ORN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Aynur KOYUNCU, Principal Investigator, Assist Prof, Hasan Kalyoncu University
Other Study IDs: HasanKUUU
Record Dates: First submitted 2023-01-11; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Work-Related Condition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Operation Room Nurses
  Interventions: Other: the operating room environment risk

INTERVENTIONS:
Other: the operating room environment risk — in determining the risks they face in the operating room environment.

SUMMARY:
Operating Room Nurses (ORN) are exposed to a lot of risks related to the working environment. There is a limited number of studies describing the risks faced by ADs in the work environment.

Aims: In this study, we aimed to determine the risk factors faced by AHs in operating rooms.

DETAILED DESCRIPTION:
Background: Operating Room Nurses (AH) are exposed to a lot of risks related to the working environment. There is a limited number of studies describing the risks faced by ADs in the work environment.

Aims: In this study, we aimed to determine the risk factors faced by AHs in operating rooms.

Study Design: This is a prospective descriptive study. Methods: The study was carried out with the operating room nurses working in the operating rooms of six hospitals affiliated to the General Secretariat of the Gaziantep Provincial Public Hospitals Association between September 2019 and February 2023.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer nurse
* Being an operating room nurse

Exclusion Criteria:

• Nurses working outside the operating room

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Being an operating room nurse
Sampling Method: Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-21 (Estimated)

PRIMARY OUTCOMES:
Determining the exposure of ORNs to radiation, biological, ergonomic, chemical, psychological and physical risks in the working environment. | 15 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - 25 December State Hospital, Gaziantep
  - Gaziantep University Şahinbey Research and Application Hospital, Gaziantep, Şahinbey

IPD SHARING:
Plan to Share IPD: Undecided